CLINICAL TRIAL: NCT03109015
Title: Alternative Schedule Sunitinib in Metastatic Renal Cell Carcinoma: Cardiopulmonary Exercise Testing
Acronym: ASSET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00072588
Record Dates: First submitted 2017-04-06; First posted 2017-04-11 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Carcinoma, Renal Cell
Keywords: metastatic renal cell carcinoma; sunitinib; Sutent; cardiopulmonary function
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Schedule 4/2 (Active Comparator)
  Interventions: Drug: Sunitinib
- Schedule 2/1 (Experimental)
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Patients randomized to sunitinib schedule 4/2 will receive sunitinib at 50 mg daily for 4 weeks on, followed by 2 weeks off, per standard of care. Cardiopulmonary Exercise Testing (CPET) will be performed at baseline, 4 weeks and 12 weeks.
  Other Names: Sutent
  Arms: Schedule 4/2
Drug: Sunitinib — Patients randomized to sunitinib schedule 2/1 will receive sunitinib 50 mg daily for 2 weeks on, followed by 1 week off. Cardiopulmonary Exercise Testing (CPET) will be performed at baseline, 5 weeks and 12 weeks.
  Other Names: Sutent
  Arms: Schedule 2/1

SUMMARY:
The purpose of this study is to determine the effect of a sunitinib administration schedule 2/1 (2 weeks of treatment followed by 1 week without) compared to a schedule 4/2 (4 weeks of treatment followed by 2 weeks without) on cardiopulmonary function in subjects with renal cell carcinoma. Subjects will be randomized 1:1 to one of two arms: 4/2 schedule of sunitinib administration or 2/1 schedule of sunitinib administration. Cardiopulmonary function will be assessed at baseline, week 4 (4/2 schedule only), week 5 (2/1 schedule only) and week 12. The investigators hypothesize that schedule 2/1 of sunitinib is not only better tolerated but will be associated with less fatigue and functional cardiovascular/muscular toxicity than the 4/2 schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histologically confirmed renal cell carcinoma (RCC)
3. One of the two following populations:

   1. High risk for recurrence of RCC after nephrectomy, in the opinion of the investigator, OR
   2. Locally advanced, unresectable or metastatic disease, in the opinion of the investigator, and good or intermediate risk by IDMC Heng Criteria (see Appendix I).
4. Karnofsky Performance Status (KPS) ≥ 80 (see Appendix A)
5. Good or intermediate risk by IDMC Heng Criteria (see Appendix I).4
6. Appropriate for treatment with sunitinib in the opinion of the treating physician.
7. Able to swallow sunitinib and comply with study requirements.
8. Able to walk and jog on a treadmill, in the opinion of the treating physician.
9. Must be able to complete an acceptable cardiopulmonary exercise test (CPET) at baseline (see Section 8.2), defined as at least one of the following:

   * Achieving a plateau in oxygen consumption concurrent with an increase in power output;
   * Respiratory exchange ratio ≥ 1.1 (RER);
   * Volitional exhaustion with a rating of perceived exertion ≥17 (RPE).
10. Subjects must have normal organ and marrow function as defined below:

    * Absolute neutrophil count ≥1,200/µL
    * Hemoglobin ≥9 g/dL
    * Platelets ≥75,000/µL
    * Total bilirubin ≤1.5 x institutional upper limit of normal
    * AST(SGOT)/ALT(SGPT) <2.5 x institutional upper limit of normal
    * Urine protein creatinine (UPC) ratio of <1 (see Appendix G schedule of events footnote)
    * Creatinine ≤2.0 OR creatinine clearance >30 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal (see Appendix H).
    * Left ventricular ejection fraction (LVEF) ≥lower limit of institutional normal as assessed by echocardiography.
11. For the sixteen patients who elect to participate in the optional technology portion involving electronic step counts and blood pressure monitoring, the patient must have a Bluetooth-enabled smart phone, which is compatible with the wireless health monitors.
12. For women of childbearing potential (WOCBP) must have a negative serum pregnancy test prior to the start of the study. Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of the study. Medically acceptable contraceptives include: (1) surgical sterilization (such as a tubal ligation or hysterectomy), (2) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (3) barrier methods (such as a condom or diaphragm) used with a spermicide, or (4) an intrauterine device (IUD). Contraceptive measures such as Plan B (TM), sold for emergency use after unprotected sex, are not acceptable methods for routine use. If you do become pregnant during this study or if you have unprotected sex, you must inform your study physician immediately.
13. For men who are sexually active, must agree to use a two medically acceptable forms of birth control (one of which must include a condom as a barrier method of contraception) in order to be in this study. Medically acceptable contraceptives include: (1) surgical sterilization (such as a vasectomy), or (2) a condom used with a spermicide. Contraceptive measures such as Plan B (TM), sold for emergency use after unprotected sex, are not acceptable methods for routine use. Men must also agree to inform their partner of the potential for harm to an unborn child. She should know that if pregnancy occurs, the subject will need to report it to the study doctor, and she should promptly notify her doctor. The study doctor will ask if the subject's partner is willing to provide updates on the progress of the pregnancy and its outcome. If the subject's partner agrees, this information will be provided to Pfizer, Inc. for safety monitoring follow-up.

Exclusion Criteria:

1. Any prior anti-VEGF therapies (i.e., sunitinib, sorafenib, pazopanib, axitinib, cabozantinib, bevacizumab, etc.), including in the adjuvant or neoadjuvant setting.
2. Prior systemic therapy for advanced RCC; however, treatment with immunotherapy (i.e., high-dose bolus IL-2, ipilimumab + nivolumab, etc.) is allowed.
3. Subjects who are receiving any other investigational agents.
4. Subjects who are receiving strong CYP3A4 inhibitors or CYP3A4 inducers (see Section 5.3.2.2).
5. Radiotherapy within 2 weeks prior to taking the first dose of study drug, or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier.
6. Central nervous system (CNS) metastases at baseline, with the exception of those subjects who have previously treated CNS metastases (surgery ± radiotherapy, radiosurgery, or gamma knife) and who meet both of the following criteria: a) are asymptomatic, and b) have no requirement for steroids or enzyme-inducing anticonvulsants in the prior 28 days.
7. Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

   * Active peptic ulcer disease
   * Known intraluminal metastatic lesion(s) with risk of bleeding
   * Inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease) or other gastrointestinal conditions with increased risk of perforation
   * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment
8. History of any one or more of the following cardiovascular conditions within the past 6 months:

   * Cardiac angioplasty or stenting
   * Myocardial infarction
   * Unstable angina
   * Coronary artery bypass graft surgery
   * Symptomatic peripheral vascular disease
   * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA) (see Appendix J)
9. Absolute contraindications to cardiopulmonary exercise testing and/or aerobic training, as determined by the attending oncologist:

   Absolute Contraindications
   * Uncontrolled arrhythmia causing symptoms or hemodynamic compromise
   * Recurrent syncope
   * Active endocarditis
   * Acute myocarditis or pericarditis
   * Symptomatic severe aortic stenosis
   * Uncontrolled heart failure
   * Suspected dissecting aneurysm
   * Uncontrolled asthma
   * Pulmonary edema
   * Room air desaturation at rest <85%
   * Respiratory failure
   * Acute non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (i.e., infection, renal failure, thyrotoxicosis)
   * Mental impairment leading to inability to cooperate.
10. Poorly controlled hypertension [defined as systolic blood pressure (SBP) of >150 mmHg or diastolic blood pressure (DBP) of >90 mmHg].
11. History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism, or untreated deep venous thrombosis (DVT) within the past 6 months.
12. Major surgery or trauma within 28 days prior to first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement are not considered to be major surgery).
13. Osseous metastatic disease with unacceptable risk of impending fracture due to study assessments, in the opinion of the investigator
14. Evidence of active bleeding or bleeding diathesis.
15. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harrison, MD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Schedule 4/2 | Schedule 2/1
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Schedule 4/2 | Schedule 2/1 | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Median (Full Range); unit: years] | 59 [52 to 66] | 68 [65 to 76] | 65 [52 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 31.27 [30.09 to 37.52] | 26.55 [15.98 to 30.58] | 30.53 [15.98 to 37.52]

OUTCOME MEASURES:

1. Primary Outcome: Change in Relative VO2 Peak From Baseline to Week 12 in the 4/2 and 2/1 Sunitinib Administration Schedules
Description: Exercise Capacity will be assessed using Cardiopulmonary Exercise Testing (CPET) to determine VO2peak. Higher VO2 peak measured in mg/ml/min indicates better cardiac function. Mean change in cardiac functions will be assessed by the difference in Relative Peak VO2 from baseline to 12 weeks in both the arms.
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Schedule 4/2 | Schedule 2/1
Number analyzed (Participants) | 4 | 3
mL/kg/min | -1.13 (2) | 1.27 (1.9)

2. Secondary Outcome: Change in Difference Between Rest Left Ventricular Ejection Fraction (LVEF) and Cardiac Function by 2-D Echocardiography (2DE) From Baseline to Week 12 in the 4/2 and 2/1 Sunitinib Administration Schedules
Description: Mean change in cardiac functions will be assessed by the difference in LVEF measured by 2D-Echo from baseline to 12 weeks in both the arms. Higher LVEF measured in percentage indicates better cardiac function.
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Schedule 4/2 | Schedule 2/1
Number analyzed (Participants) | 4 | 3
percentage | 1.5 (4.1) | -9.0 (10.6)

3. Secondary Outcome: Change in Difference Between Rest and Stress Left Ventricular Ejection Fraction (LVEF) and Cardiac Function by 3-D Echocardiography (3DE) From Baseline to Week 12 in the 4/2 and 2/1 Sunitinib Administration Schedules [Time Frame: Baseline, Week 12]
Time Frame: Baseline, week 12
Population: No data collected
Arm/Group | Schedule 4/2 | Schedule 2/1
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in One Repetition Maximum (1RM) in Upper and Lower Extremity Muscular Strength From Baseline to Week 12 in the 4/2 and 2/1 Sunitinib Administration Schedules
Description: Mean change in upper and lower extremity maximal muscular strength as measured by the voluntary one-repetition max (1-RM) between week 12 and baseline. A 1-RM is defined as the greatest resistance that can be moved through the full range of motion in a controlled manner. This assessment included following exercises: leg press, chest press, and row. The heaviest weight lifted while adhering to the strict technique and form will be used to score the assessment.
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Schedule 4/2 | Schedule 2/1
Number analyzed (Participants) | 4 | 3
pounds
  Seated Row | 7 (20) | 6.67 (35.2)
  Chest Press | -6.5 (12.7) | -6.0 (18.5)
  Leg Press | 52.25 (83.1) | 15 (105)

5. Secondary Outcome: Change in Muscular Endurance in Upper and Lower Extremity Muscular Strength From Baseline to Week 12 in the 4/2 and 2/1 Sunitinib Administration Schedules
Description: Mean change in upper and lower extremity maximal muscular strength as measured by the muscular endurance which is 70% of 1-RM between week 12 and baseline. Muscular Endurance of the upper and lower body will be assessed as the number of repetitions to fatigue at 70% of the 1-RM. The same exercises and methods will be used as in the 1-RM determination.
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Schedule 4/2 | Schedule 2/1
Number analyzed (Participants) | 4 | 3
pounds
  Seated Row | 1.25 (7.5) | 4.33 (24.8)
  Chest Press | -4.5 (8.9) | -4.0 (12.5)
  Leg Press | 36.5 (58.9) | 10.33 (73.5)

6. Secondary Outcome: Change in Muscle Cross-sectional Area (CSA) of the Major Muscles Near Lumbar3 (CT Scans and Slice-O-Matic® Software) From Baseline to Week 12 in the 4/2 and 2/1 Sunitinib Administration Schedules [Time Frame: Baseline, Week 12]
Time Frame: Baseline, week 12
Population: No data collected
Arm/Group | Schedule 4/2 | Schedule 2/1
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Time Taken to Complete the 5-repititionChair-stand Test From Baseline to Week 12 in the 4/2 and 2/1 Sunitinib Administration Schedules
Description: The 5-repetition Chair-Stand Test measures the time taken to complete 5 repetitions of the sit-to-stand maneuver performed on a chair. Standardized instructions are: "By the count of 3, please stand up and sit down as quickly as possible for 5 times. Place your hands on your lap, and do not use them throughout the procedure. Lean your back against the chair's backrest at the end of every repetition." Note: Timing will start when the subject's back left the backrest and will be stopped once the back touched the backrest.
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Schedule 4/2 | Schedule 2/1
Number analyzed (Participants) | 4 | 3
seconds | -0.43 (0.9) | -2.05 (0.5)

8. Secondary Outcome: Change in Time Taken to Complete the Timed up and Go Test From Baseline to Week 12 in the 4/2 and 2/1 Sunitinib Administration Schedules
Description: Timed Up and Go (TUG) test assesses a person's mobility. TUG measures the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. Scores of 10 seconds or less indicate normal mobility, 11 - 20 seconds are within normal limits for frail, elderly, and disabled subjects, and greater than 20 seconds suggests that further examination is required.
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Schedule 4/2 | Schedule 2/1
Number analyzed (Participants) | 4 | 3
seconds | -0.5 (1.3) | 0 (1.7)

9. Secondary Outcome: Change in Distance Walked During the 6 Minute Walk Test From Baseline to Week 12 in the 4/2 and 2/1 Sunitinib Administration Schedules
Description: Subjects will be instructed to cover the longest distance possible in 6 minutes under the supervision of an exercise physiologist or trained designee. The walked distance will be determined in a measured corridor between 2 cones that were placed 30 meters apart
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Schedule 4/2 | Schedule 2/1
Number analyzed (Participants) | 4 | 3
meters | 1.43 (13.3) | -69.2 (83.1)

10. Secondary Outcome: Change in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Scale Score From Baseline to Week 12 in the 4/2 and 2/1 Sunitinib Administration Schedules
Description: Mean change in PRO: FACIT-Fatigue (FACIT-F, range 0 to 52) aggregate score between week 12 and baseline. Higher scores indicate better quality of life.
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Schedule 4/2 | Schedule 2/1
Number analyzed (Participants) | 4 | 3
score on a scale | -2.89 (3.8) | -2.87 (5.2)

11. Secondary Outcome: Change in Functional Assessment of Cancer Therapy - Kidney Symptom Index - 19 (FKSI-19) Score From Baseline to Week 12 in the 4/2 and 2/1 Sunitinib Administration Schedules
Description: Mean change in PRO: FKSI- 19 (FKSI-19 Range 0 to 76) aggregate score between week 12 and baseline. Higher scores indicate better quality of life.
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Schedule 4/2 | Schedule 2/1
Number analyzed (Participants) | 4 | 3
score on a scale | 2.75 (4.8) | -1.0 (3.6)

12. Secondary Outcome: Change in Hospital Anxiety and Depression Survey (HADS) Score From Baseline to Week 12 in the 4/2 and 2/1 Sunitinib Administration Schedules
Description: Mean change in PRO: HADS (HADS, range 0 to 21) aggregate score between week 12 and baseline. The HADS score has 2- subscales: Depression and Anxiety. Each sub-scale ranges from 0, 21. Higher scores indicate higher levels of depression and anxiety.
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Schedule 4/2 | Schedule 2/1
Number analyzed (Participants) | 4 | 3
score on a scale
  Change in Anxiety (HADS) | 0.75 (1.5) | 0.3 (1.1)
  Change in Depression (HADS) | 0.0 (2.4) | 1.3 (2.9)

13. Secondary Outcome: Change in Leisure Activity Score From the Godin-Leisure Questionnaire From Baseline to Week 12 in the 4/2 and 2/1 Sunitinib Administration Schedules
Description: Mean change in PRO: Godin-Leisure questionnaire aggregate score between week 12 and baseline. This represents the activity level of a participant. There are no standard reference range for this assessment. Higher scores indicate higher physical activity.
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Schedule 4/2 | Schedule 2/1
Number analyzed (Participants) | 4 | 3
score on a scale | 1.67 (17.6) | 0.5 (36.1)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Schedule 4/2 | Schedule 2/1
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Schedule 4/2 (N=4) | Schedule 2/1 (N=3)
Fatigue (General disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Schedule 4/2 (N=4) | Schedule 2/1 (N=3)
Neutrophil count decreased (Investigations) | 0 | 1
Weight loss (Investigations) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Blurred vision (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Hypogeusia (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 3 | 3
Flu like symptoms (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Cellulitis, left knee (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Gout, left knee (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1
Hypertension (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT03109015/Prot_SAP_000.pdf